CLINICAL TRIAL: NCT01543867
Title: Non-interventional Study of the Safety and Efficacy of Long-term Somatropin Treatment in Children (GrowthWIN II / GrowthWIN II SGA)
Brief Title: Safety and Efficacy of Long-term Somatropin Treatment in Children
Acronym: GrowthWIN II
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-1930
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children; Foetal Growth Problem; Small for Gestational Age; Genetic Disorder; Turner Syndrome; Growth Disorder; Idiopathic Short Stature
MeSH Terms: conditions — Genetic Diseases, Inborn; Turner Syndrome; Growth Disorders | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Users of somatropin
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Prescribed at the discretion of the treating physician according to product labelling

SUMMARY:
This study is conducted in Europe. The aim of this study is to evaluate safety during the long-term use of somatropin (Norditropin®) in children as well as efficacy on change in height. A subgroup of children small for their gestational age is included.

ELIGIBILITY:
Inclusion Criteria:

* In need of somatropin or current user

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children treated with somatropin
Sampling Method: Probability Sample
Enrollment: 5442 (Actual)
Dates: Start 2001-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Up to 10 years

SECONDARY OUTCOMES:
Number of patients continuing somatropin treatment | Up to 10 years
Change in height | Up to 10 years
Onset of puberty in children small for gestational age | Up to 10 years
Co-morbidities in children small for gestational age | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Mainz, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com